CLINICAL TRIAL: NCT02520518
Title: Does Dapagliflozin Promote Favorable Health Benefits That Are Independent Of Weight Loss?
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Designed a new modified/simplified protocol see NCT 03180489
Sponsor: Christopher Bell (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-5531H
Record Dates: First submitted 2015-07-27; First posted 2015-08-13 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — dapagliflozin; Body Weight Maintenance; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dapagliflozin: ad libitum dietary intake (Experimental): Daily oral administration of dapagliflozin with ad libitum dietary intake. The dose of dapagliflozin will begin as one 5 mg tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two 5 mg tablets per day for the remainder of the study.
  Interventions: Drug: Dapagliflozin; Behavioral: Ad libitum dietary intake
- Dapagliflozin: weight maintenance (Experimental): Daily oral administration of dapagliflozin with supplemented dietary intake to achieve weight maintenance. The dose of dapagliflozin will begin as one 5 mg tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two 5 mg tablets per day for the remainder of the study.
  Interventions: Drug: Dapagliflozin; Behavioral: Weight maintenance
- Placebo: ad libitum dietary intake (Placebo Comparator): Daily oral administration of a placebo with ad-libitum dietary intake. Matching placebo for dapagliflozin 5 mg will begin as one tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two tablets for the remainder of the study.
  Interventions: Drug: Placebo; Behavioral: Ad libitum dietary intake
- Placebo: dietary restriction (Placebo Comparator): Daily oral administration of a placebo plus dietary restriction such that weight loss is matched to participants in Arm 1. Matching placebo for dapagliflozin 5 mg will begin as one tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two tablets for the remainder of the study.
  Interventions: Drug: Placebo; Behavioral: Dietary restriction

INTERVENTIONS:
Drug: Dapagliflozin
  Other Names: Farxiga
  Arms: Dapagliflozin: ad libitum dietary intake; Dapagliflozin: weight maintenance
Drug: Placebo
  Arms: Placebo: ad libitum dietary intake; Placebo: dietary restriction
Behavioral: Weight maintenance
  Arms: Dapagliflozin: weight maintenance
Behavioral: Ad libitum dietary intake
  Arms: Dapagliflozin: ad libitum dietary intake; Placebo: ad libitum dietary intake
Behavioral: Dietary restriction
  Arms: Placebo: dietary restriction

SUMMARY:
Th mechanism of action of dapagliflozin is via sodium-glucose co-transporter 2 (SGLT2) inhibition. Sodium-glucose co-transporter 2 inhibition is associated with moderate weight (fat) loss, in addition to other health benefits, including decreased blood pressure, decreased inflammation, and decreased oxidative stress. It is unclear as to whether these health benefits are due to SGLT2 inhibition per se, or as a secondary effect of weight loss.

DETAILED DESCRIPTION:
This is a randomized, prospective, placebo-controlled, double-blind, repeated measures study. 92 overweight/obese adults (body mas index > 27.5 kg/m^2) will be recruited for participation and randomly assigned to one of four 12 week treatments: 1) daily oral administration of dapagliflozin with ad-libitum dietary intake; 2) daily oral administration of dapagliflozin with supplemented dietary intake to achieve weight maintenance; 3) daily oral administration of a placebo plus dietary restriction such that weight loss is matched to participants in treatment 1; or, 4) daily oral administration of a placebo with ad-libitum dietary intake.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Aged 18-65 years.
3. No known Type 2 Diabetes
4. Body mass index greater than or equal to 27.5 kg/m^2
5. Sedentary (maximum of 2/week regularly scheduled activity sessions of < 20 minutes during the previous 2 years)
6. Completion of a screening visit consisting of medical history, physical examination, and 12-lead electrocardiogram and blood pressure assessment at rest and during incremental exercise to volitional exhaustion (Note: Subjects with abnormal screening values may be eligible if the results are not clinically significant, as judged by the investigator or medical monitor)
7. Agree to abide by the study schedule and dietary restrictions and to return for the required assessments
8. Women of childbearing potential must have negative pregnancy test and be using acceptable contraception

Exclusion Criteria:

1. Evidence of clinically significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, haematological, neurological, psychiatric, or other disease that may interfere with the objectives of the study or the safety of the subject, as judged by the investigator in agreement with the sponsor or medical monitor, have been hospitalized in the past 2 years as a result of these conditions, or are receiving pharmacological treatment for these conditions
2. Use of prescription drugs (see exceptions listed below) or herbal preparations in the 4 weeks before study commencement.

   Permitted Prescription Drugs
   * Birth Control
   * Less than 7 days, short course antibiotics. Note: Rifampin is not permitted.
   * Other medicines, for Gastroesophageal Reflux Disease (GERD), depression, seasonal allergies and over-the-counter analgesics, maybe allowed, but will be approved on a case-by-case basis.
3. Is currently enrolled in another clinical study for another investigational drug or has taken any other investigational drug within 30 days before the screening visit.
4. Habitual and/or recent use (within 2 years) of tobacco
5. Being considered unsuitable for participation in this trial for any reason, as judged by the investigator or medical monitor.
6. History of serious hypersensitivity reaction to dapagliflozin
7. Severe renal impairment, end-stage renal disease, or dialysis
8. Pregnant or breastfeeding patients
9. Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal and/or alanine aminotransferase (ALT) >3x upper limit of normal
10. Total bilirubin >2.0 mg/dL (34.2 umol/L)
11. Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody Immunoglobulin M, Hepatitis B surface antigen and Hepatitis C virus antibody
12. Estimated Glomerular Filtration Rate <60 mL/min/1.73 m^2 (calculated by Cockcroft-Gault formula).
13. History of bladder cancer
14. Recent cardiovascular events in a patient, including any of the following: acute coronary syndrome within 2 months prior to enrollment; hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrollment; acute stroke or trans-ischemic attack within two months prior to enrollment; less than two months post coronary artery revascularization; congestive heart failure defined as New York Heart Association class IV,unstable or acute congestive heart failure. Note: eligible patients with congestive heart failure, especially those who are on diuretic therapy, should have careful monitoring of their volume status throughout the study
15. Blood pressure at enrolment: Systolic blood pressure ≥165 mmHg and/or diastolic blood pressure ≥100 mmHg
16. Blood pressure at randomization: Systolic blood pressure ≥165 mmHg and/or diastolic blood pressure ≥100 mmHg
17. Patients who, in the judgment of the medical monitor, may be at risk for dehydration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin: ad Libitum Dietary Intake: Daily oral administration of dapagliflozin with ad libitum dietary intake. The dose of dapagliflozin will begin as one 5 mg tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two 5 mg tablets per day for the remainder of the study.
  Dapagliflozin
  Ad libitum dietary intake
- Dapagliflozin: Weight Maintenance: Daily oral administration of dapagliflozin with supplemented dietary intake to achieve weight maintenance. The dose of dapagliflozin will begin as one 5 mg tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two 5 mg tablets per day for the remainder of the study.
  Dapagliflozin
  Weight maintenance
- Placebo: ad Libitum Dietary Intake: Daily oral administration of a placebo with ad-libitum dietary intake. Matching placebo for dapagliflozin 5 mg will begin as one tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two tablets for the remainder of the study.
  Placebo
  Ad libitum dietary intake
- Placebo: Dietary Restriction: Daily oral administration of a placebo plus dietary restriction such that weight loss is matched to participants in Arm 1. Matching placebo for dapagliflozin 5 mg will begin as one tablet per day for the first 14-days. In the absence of complications, side effects, or unfavorable reactions, the dose will then increase to two tablets for the remainder of the study.
  Placebo
  Dietary restriction
Period: Overall Study
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Started | 3 | 1 | 3 | 2
Completed | 3 | 1 | 1 | 1
Not Completed | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Some of the participants with baseline measures collected either declined participation or were enrolled in the amended protocol NCT03180489.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction | Total
Number analyzed (Participants) | 3 | 1 | 3 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 3 | 2 | 9
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 2 | 9
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 3 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Sensitivity at Week 12
Description: Via oral glucose tolerance test.
Time Frame: Baseline,12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Blood Pressure at Week 12
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: Dietary Restriction | Placebo: ad Libitum Dietary Intake
Number analyzed (Participants) | 3 | 1 | 2 | 3
mmHg
  Systolic Blood Pressure Change | 2 (1) | 5 (0) | 11 (8) | 0 (3)
  Diastolic Blood Pressure Change | -1 (0.2) | -1 (0) | 11 (4) | 1 (2)

3. Primary Outcome: Change From Baseline in Perception of Satiety at Week 12
Description: Perceptions of satiety will be determined using a visual analog scale called a Hunger Rating Scales. The minimum value is 1 (not at all full) and the maximum value is 100 (extremely full). One value between 1 and 100 is reported by the participant dependent on their perception. No sub scores are used. The perceived values are reported as the group average at baseline and 12 weeks. There is not a better or worse outcome, but rather a measure of perceived satiety. If Dapagliflozin were effective at increasing fullness, respondents would exhibit 12-week scores for the question in comparison to their baseline scores.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: Dietary Restriction | Placebo: ad Libitum Dietary Intake
Number analyzed (Participants) | 3 | 1 | 1 | 3
score on a scale
  Baseline | 50 (14) | 61 (0) | 35 (34) | 39 (14)
  12 weeks | 56 (29) | 33 (0) | 38 (0) | 42 (10)

4. Primary Outcome: Change From Baseline in Perception of Hunger at Week 12
Description: Perceptions of Hunger will be determined using a visual analog scale called a Hunger Rating Scales. The minimum value is 1 (not at all hungry) and the maximum value is 100 (very hungry). One value between 1 and 100 is reported by the participant dependent on their perception. No sub scores are used. The perceived values are reported as the group average at baseline and 12 weeks. There is not a better or worse outcome, but rather a measure of perceived hunger. If Dapagliflozin were effective at decreasing hunger, respondents would exhibit 12-week scores for the question in comparison to their baseline scores.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: Dietary Restriction | Placebo: ad Libitum Dietary Intake
Number analyzed (Participants) | 3 | 1 | 1 | 3
score on a scale
  Baseline | 20 (22) | 24 (0) | 23.5 (1) | 32 (27)
  12 weeks | 28 (38) | 77 (0) | 65 (0) | 31 (15)

5. Primary Outcome: Change From Baseline in Marker of Inflammation (High Sensitive C-reactive Protein) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: Change From Baseline in Marker of Inflammation (Tumor Necrosis Factor Alpha) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data collection was not performed
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Primary Outcome: Change From Baseline in Marker of Inflammation (Interleukin 6) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data collection was not performed
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Primary Outcome: Change From Baseline in Hunger Hormone Ghrelin at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Primary Outcome: Change From Baseline in Hunger Hormone Peptide Tyrosine Tyrosine at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Primary Outcome: Change From Baseline in Maker of Oxidative Stress (Oxidized Low Density Lipoprotein) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Primary Outcome: Change From Baseline in Maker of Oxidative Stress (Low Density Thiobarbituric Acid Reactive Substances) at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Primary Outcome: Change From Baseline in Satiety Hormone Leptin at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Primary Outcome: Change From Baseline in Satiety Hormone Insulin at Week 12
Description: Will be analyzed using a commercially available biochemical assay.
Time Frame: Baseline, 12 weeks
Population: Data were not collected.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: During the 12 week intervention period
Description: This study was performed on a healthy population and mortality is not an outcome. All cause mortality was monitored.
Arm/Group | Dapagliflozin: ad Libitum Dietary Intake | Dapagliflozin: Weight Maintenance | Placebo: ad Libitum Dietary Intake | Placebo: Dietary Restriction
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 1/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin: ad Libitum Dietary Intake (N=3) | Dapagliflozin: Weight Maintenance (N=1) | Placebo: ad Libitum Dietary Intake (N=3) | Placebo: Dietary Restriction (N=2)
Stomach Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loose Stool (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
increase in urination (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever and sore throat (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stuffy Nose (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02520518/Prot_SAP_ICF_000.pdf